CLINICAL TRIAL: NCT06727526
Title: The Effect of Acupressure on Pain and Physiological Parameters in Infants Before and After Cardiac Catheterization: a Randomized Placebo Controlled Trial
Brief Title: Acupressure's Impact on Pain and Physiological Parameters in Infants Undergoing Cardiac Catheterization
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Baskent University (Other)
Responsible Party: Principal Investigator, Ilcim Ercan Koyuncu, Principal Investigator, Istanbul University - Cerrahpasa
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: Acupressure in Infants
Record Dates: First submitted 2024-12-09; First posted 2024-12-11 (Actual); Last update posted 2024-12-17 (Actual); Status verified 2024-12

CONDITIONS: Cardiac Catheterization
Keywords: cardiac catheterization; congenital heart disease; Acupressure; nursing care; pain
MeSH Terms: conditions — Heart Defects, Congenital; Pain | interventions — Acupressure

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Acupressure Group (Experimental): Infants in this group will undergo acupressure both before and after cardiac catheterization. The initial session will be administered by the researcher 30 minutes prior to the procedure. Acupressure will target three specific points: the seventh point of the heart meridian (HT7), the fourth point of the large intestine meridian (LI4), and the sixth point of the pericardial meridian (PC6). The areas will be warmed for approximately 20 seconds to minimize tissue sensitivity, avoiding direct pressure on the acupressure points. Each point will receive 12 minutes of treatment, comprising 10 seconds of compression followed by 2 seconds of relaxation, applied symmetrically. After this initial session, the infant will undergo cardiac catheterization. Upon return to the ward post-catheterization, a second acupressure session will be conducted one hour after the administration of the final dose of ketamine hydrochloride.
  Interventions: Other: Acupressure
- Plasebo (Placebo Comparator): Infants in this group will receive placebo acupressure before and after cardiac catheterization. The initial session will be administered 30 minutes before the procedure, targeting areas approximately 1-1.5 cm away from HT7, LI4, and PC6 points, where meridians do not pass. The areas will be warmed for 20 seconds to minimize tissue sensitivity, avoiding direct pressure on acupressure points. Each site will receive 12 minutes of treatment, alternating 10 seconds of compression and 2 seconds of relaxation, applied symmetrically. Post-catheterization, a second placebo session will be conducted an hour after the last dose of ketamine hydrochloride.
  Interventions: Other: Placebo acupressure
- Control Group (No Intervention): Infants in this group will not receive any specific intervention and will be provided routine care in the ward.

INTERVENTIONS:
Other: Acupressure — The literature found that acupressure positively affects child health, but no study was found to determine the effect of acupressure on pain and physiological parameters in children undergoing cardiac catheterization. Therefore, this study was designed to determine the effect of acupressure applied before and after cardiac catheterization on infants' pain levels and physiological parameters.
  Arms: Acupressure Group
Other: Placebo acupressure — In health sciences, placebo refers to an inactive intervention used to relax the patient and assess treatment efficacy. It may involve inert substances (e.g., sugar tablets, saline) or non-therapeutic interventions (e.g., artificial electrical stimulation or conversations). Expectancy theory often explains The placebo effect, which suggests that treatment expectations can induce physiological changes. Factors like age, cognitive development, and previous pain experiences influence children's responses to placebo. Parental belief in an intervention's efficacy can reduce a child's pain expectations and positively influence their perception of pain. Although the sample included young children, our study incorporated the placebo group to account for this effect, especially since the parents evaluated pain scores.
  Arms: Plasebo

SUMMARY:
Acupressure, one of the traditional Chinese medicine practices dating back approximately 5,000 years, is a mind-body technique that can be independently applied by nurses. This practice involves applying pressure to specific points on the body to reduce pain. The pressure stimulates the release of substances such as endorphins, acetylcholine, norepinephrine, and dopamine, resulting in muscle relaxation, regulated blood circulation, and blocked pain signals at nerve endings, effectively reducing the sensation of pain. The aim of acupressure is to alleviate patient discomfort and improve quality of life by reducing the need for analgesics. Acupressure, which falls under the category of therapeutic massage, can be applied using the fingers and palms. According to its core philosophy, illness arises when the balance of energy flowing through body channels, called "meridians," is disrupted. Because acupressure does not involve needles, it is a safe, effective, and economical technique that is easy to learn and apply. The World Health Organization (WHO) classifies acupressure as a supportive treatment within its list of "treatable conditions." The technique involves applying pressure to the same point for 2-5 minutes. Stimulating specific points promotes the release of cytokines, such as endorphins, which play a role in pain reduction by blocking certain receptors on sensory nerve endings and thus preventing pain perception. Additionally, stimulating acupoints helps establish sympathetic and parasympathetic balance, supporting healthy homeostasis. Studies in the literature have investigated acupressure's positive effects on children's preoperative anxiety, postoperative pain severity, chemotherapy side effects, fatigue, sleep quality, asthma symptoms, and physical stress. In a study examining the impact of acupressure on procedural pain in infants prior to parenteral vaccinations, infants who received acupressure experienced lower pain levels and shorter crying durations. Similarly, a study investigating the effect of acupressure on acute pain during venous catheter insertion in children found that pain severity was lower among children who received acupressure. A systematic review examining the effects of acupressure on child health determined that acupressure is effective in alleviating procedural pain in children. The review emphasized that nurses should incorporate acupressure, a non-pharmacological method, into care practices for effective pain management in children. Despite evidence in the literature supporting acupressure's positive effects on pediatric health, no study has specifically examined its impact on pain and physiological parameters in children undergoing cardiac catheterization. Therefore, this thesis aims to investigate the effects of acupressure, applied before and after cardiac catheterization, on pain levels and physiological parameters in infants.

ELIGIBILITY:
Inclusion Criteria:

* Infants between 1 month and 12 months
* Infants with congenital heart disease
* Infants undergoing cardiac catheterization for the first time
* Infants undergoing planned cardiac catheterization
* Infants without acupressure experience
* Infants whose parents volunteered to participate in the study

Exclusion Criteria:

* Infants with complications during catheterization
* Infants followed up in the intensive care unit after catheterization
* Infants with any deformity or lesion in the acupressure area
* Infants who have not received analgesics after catheterization
* Infants who were not given analgesics within six hours before catheterization
* Infants with neurodevelopmental disorders
* Infants whose parents did not volunteer to participate in the study

Ages: 1 Month to 12 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 35 (Estimated)
Dates: Start 2024-12-30 (Estimated); Primary Completion 2024-12-31 (Estimated); Study Completion 2025-12-30 (Estimated)

PRIMARY OUTCOMES:
Pain | 30 minutes after the first procedure, 30 minutes after the second procedure, 2 hours after the second procedure, 24 hours after the second procedure
  The Face, Legs, Activity, Cry, Consolability (FLACC) scale will assess the pain. The FLACC scale is a measurement used to assess pain for children between the ages of 1 month and 7 years or individuals who are unable to communicate their pain. The scale is scored in a range of 0-10, with 0 representing no pain. As the score increases, the patient's pain increases.

SECONDARY OUTCOMES:
Heart Rate | 30 minutes after the first procedure, 30 minutes after the second procedure, 2 hours after the second procedure, 24 hours after the second procedure
  Maintaining or normalizing heart rate within normal range (100-160)
Saturation | 30 minutes after the first procedure, 30 minutes after the second procedure, 2 hours after the second procedure, 24 hours after the second procedure
  Normalizing or maintaining saturation rate within the normal range according to the child.

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Koc Ozkan T, Balci S. The Effect of Acupressure on Acute Pain During Venipuncture in Children: Implications for Evidence-Based Practice. Worldviews Evid Based Nurs. 2020 Jun;17(3):221-228. doi: 10.1111/wvn.12437. Epub 2020 Apr 22. PMID 32320139
- [Background] Bastani F, Khosravi M, Borimnejad L, Arbabi N. The effect of acupressure on cancer-related fatigue among school-aged children with acute lymphoblastic leukemia. Iran J Nurs Midwifery Res. 2015 Sep-Oct;20(5):545-51. doi: 10.4103/1735-9066.164508. PMID 26457090
- [Background] American Academy of Pediatrics, Committee on Pediatric Emergency Medicine; American College of Emergency Physicians, Pediatric Committee; Emergency Nurses Association, Pediatric Committee. Joint policy statement--guidelines for care of children in the emergency department. J Emerg Nurs. 2013 Mar;39(2):116-31. doi: 10.1016/j.jen.2013.01.003. PMID 23498882
- [Background] Alakhfash AA, Jelly A, Almesned A, Alqwaiee A, Almutairi M, Salah S, Hasan M, Almuhaya M, Alnajjar A, Mofeed M, Nasser B. Cardiac Catheterisation Interventions in Neonates and Infants Less Than Three Months. J Saudi Heart Assoc. 2020 May 12;32(2):149-156. doi: 10.37616/2212-5043.1051. eCollection 2020. PMID 33154909